CLINICAL TRIAL: NCT00754013
Title: A 10-Week, Double-Blind, Placebo-Controlled Study To Evaluate The Efficacy And Safety Of Donepezil Hydrochloride (Aricept) In The Treatment Of The Cognitive Dysfunction Exhibited By Children With Down Syndrome, Aged 6 To 10
Brief Title: Evaluating The Efficacy And Safety Of Donepezil Hydrochloride (Aricept) In The Treatment Of The Cognitive Dysfunction Exhibited By Children With Down Syndrome, Aged 6 To 10
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sufficient evidence of efficacy not met.
Sponsor: Eisai Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2020-A001-336; A2501061
Record Dates: First submitted 2008-09-15; First posted 2008-09-17 (Estimated); Results first posted 2013-02-13 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2017-02

CONDITIONS: Down Syndrome; Cognitive Dysfunction
Keywords: pediatric; Down syndrome; cognitive dysfunction; Downs; Aricept; children with Down syndrome
MeSH Terms: conditions — Down Syndrome; Cognitive Dysfunction | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Donepezil (Active Comparator)
  Interventions: Drug: Aricept (Donepezil hydrochloride)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aricept (Donepezil hydrochloride) — All subjects will start with a dose of 1.25 mg/day (1.25 ml) donepezil ; dose escalations will occur every 2 weeks to a maximum of 5 mg/day (5 ml) donepezil.
  All doses will be administered orally.
  Other Names: Donepezil hydrochloride
  Arms: Donepezil
Drug: Placebo — All subjects will start with a dose of 1.25 mg/day (1.25 ml) placebo; dose escalations will occur every 2 weeks to a maximum of 5 mg/day (5 ml) placebo.
  All doses will be administered orally.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy and safety of donepezil hydrochloride (Aricept) in the treatment of cognitive dysfunction shown by children with Down syndrome, aged 6 to 10 years.

DETAILED DESCRIPTION:
This is a multinational study with sites in the US, India, Singapore, South Korea, Mexico and Chile. There will be 210 subjects (male or female) enrolled that are residing in community or facilities with a reliable caregiver that have been clinically diagnosed with Down syndrome. The assessments performed during this study will be used to evaluate skills. The study duration will be 10 weeks of double blind treatment with a total of 6 visits; 4 in office visit and 2 phone visits.

ELIGIBILITY:
Inclusion Criteria:

* Age range: Subjects 6 to 10 years of age at the screening visit; weight >= 15 kg.
* Sex distribution: both males and females.
* VABS-II/PCRF receptive sub-domain raw score of >= 25 and expressive sub-domain raw score of >= 61.
* Clinical diagnosis of Down syndrome (DS) - subjects may have free trisomy 21, Robertsonian translocations, or mosaic DS
* Naive to approved or unapproved cholinesterase inhibitors (Aricept, Exelon, Cognex, Reminyl/Razadyne, metrifonate, physostigmine) is preferred. However, prior use of these medications is allowed, provided that the medication was discontinued at least 3 months prior to screening and that it was not discontinued for lack of tolerability or efficacy or for the sole purpose of enrolling the patient in the study. The exception to this prior use is that subjects who participated in the Phase II study E2020-A001-219 (A2501059) are not eligible.
* Subjects residing in the community or in facilities that have consistent and reliable caregivers who can provide efficacy information about the subjects.
* The subjects must be expected to complete all procedures scheduled during the Screening and Baseline visits including all efficacy and safety parameters. Subjects who are verbal and able to be understood most of the time are preferred, but those who use other forms of communication, signs, symbol boards or devices to supplement his/her communication ability may be enrolled provided they meet the VABS-II/PCRF receptive and expressive score criteria mentioned above.
* Subjects must have a parent, or other reliable caregiver who agrees to accompany the subject to all clinic visits, provide information about the subject as required by the protocol, and ensure compliance with the medication schedule.
* The parent or caregiver must be a constant and reliable informant with sufficient contact with the subject to have detailed knowledge of the subject's adaptive functioning in order to be able to complete the VABS-II/PCRF accurately. The same individual should complete the form at every visit if possible.
* Subjects should be in good general health with no medical conditions that are considered both clinically significant and unstable.
* Clinical laboratory values within normal limits or abnormalities considered not clinically significant by the investigator and sponsor.
* Subjects with stable Type I (insulin-dependent) or Type II diabetes are eligible provided they are monitored regularly prior to and during the study to ensure adequate glucose control. (Adequacy of control is based on the investigator's judgment, but should be guided primarily by a glycosylated hemoglobin [hemoglobin A1c] <8.0 at screening; other information, including records of home monitoring and the screening fasting glucose may support this judgment.)
* Subjects with thyroid disease also may be included in the study provided they are euthyroid and stable on treatment for at least 1 month prior to screening.
* Subjects with a history of seizure disorder are allowed provided that they are on stable treatment for at least 3 months and have not had a seizure within the past 6 months.
* Subjects should be independent in ambulation or ambulatory aided (i.e., walker or cane, to wheelchair); vision and hearing (eyeglasses and/or hearing aid permissible) sufficient for achieving VABS-II/PCRF minimum receptive raw scores of >= 25 and expressive scores of >= 61 and for cooperating with secondary efficacy evaluations and study examinations.

Exclusion Criteria:

* Age range: Subjects <6 or >10 years at the screening visit.
* Subjects with active or clinically significant conditions that will, in the investigator's judgment, affect absorption, distribution or metabolism of the study medication (e.g., inflammatory bowel disease, gastric or duodenal ulcers or severe lactose intolerance); controlled celiac disease is allowed.
* Subjects with a known hypersensitivity to piperidine derivatives or cholinesterase inhibitors.
* Subjects currently receiving cholinesterase inhibitors or who have received them in the 3 months prior to screening or with prior use >3 months prior to screening who stopped for lack of efficacy or tolerability or simply to enroll the subject in this study. Also excluded are subjects who participated in the Phase II study E2020-A001-219 (A2501059). In addition, subjects may not have taken any other investigational medications (including memantine) within 3 months prior to screening.
* Subjects without a reliable parent or caregiver (caregiver responsibilities are described in the Inclusion Criteria above), or with parents or caregivers who are unwilling or unable to complete any of the outcome measures and fulfill the requirements of this study.
* Subjects with clinically significant obstructive pulmonary disease or asthma, untreated or not controlled by treatment within 3 months prior to screening.
* Subjects with recent (<= 1 year) or ongoing hematologic/oncologic disorders (mild anemia allowed).
* Evidence of active, clinically significant, and unstable gastrointestinal, renal, hepatic, endocrine or cardiovascular system disease.
* Subjects with a current Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) diagnosis of Major Depressive Disorder (MDD) or any current primary psychiatric diagnosis other than DS (as per DSM-IV). Diagnoses that are secondary, such as attention deficit hyperactivity disorder, are allowed.
* Any condition which would make the patient or the caregiver, in the opinion of the investigator, unsuitable for the study.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas McRae, MD, Study Director — Pfizer
Locations (2):
- United States (2):
  - Road Runner Research, San Antonio, Texas
  - NeuroScience, Inc., Herndon, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study planned to recruit subjects at 26 centers in the United States. However, the study was terminated early and only 5 centers enrolled subjects during the period of 06 Oct 2008 to 10 Dec 2008.
Groups:
- Donepezil: Donepezil was titrated to a dose of approximately 0.1-0.2 mg/kg/day as liquid containing 1 mg/1 mL of donepezil.
- Placebo: Donepezil matched placebo was titrated in the similar way as the donepezil arm.
Period: Overall Study
Arm/Group | Donepezil | Placebo
Started | 4 | 5
Completed | 0 | 0
Not Completed | 4 | 5
Not completed — Lost to Follow-up | 1 | 1
Not completed — didn't return after study termed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Donepezil | Placebo | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.0 (0.8) | 8.0 (1.4) | 8.5 (0.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 2 | 2 | 4
Race/Ethnicity, Customized [Number; unit: participants]
  White (n) | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Vineland-II Adaptive Behavior Scales (VABS-II) Parent/Caregiver Rating Form (PCRF) Sum of the 9 Sub-domain V-scores (3 Scores for Each of the Communication, Daily Living Skills, and Socialization Domains) Using Last Observation Carried Forward.
Description: The primary objective of the study was evaluation of the efficacy and safety of donepezil hydrochloride in the treatment of the cognitive dysfunction exhibited by children with Down syndrome (DS), aged 6 to 10, as assessed by analysis of VABS-II/PCRF in the domains of communication, daily living skills, and socialization, and as assessed by standard safety measurements.
Time Frame: Visit 0 (Screen), Visits 1 (Baseline), 2, and 3 (or Early Termination).
Population: The planned efficacy analysis was on the intent-to-treat (ITT) population. This study was terminated early. Primary efficacy data were not analyzed since only 9 of the 140 planned subjects had been enrolled.
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Mean Change From(Baseline) to Visit 3(Week 10 or Early Termination) in VABS-II/PCRF Sum of the 9 Sub-domain V-scores (3 Scores for Each of the Communication, Daily Living Skills, and Socialization Domains) Using Last Observation Carried Forward.
Description: The planned secondary objectives of the study included further evaluation of efficacy as assessed by additional analyses of the VABS-II/PCRF, by analyses of the Test of Verbal Expression and Reasoning (TOVER), a subject-performance-based measure of expressive language function, and by the Forward Memory and Attention Sustained sub-tests of the Leiter International Performance Scale - Revised (Leiter-R), a cognitive assessment instrument for children and adolescents that is not language dependent. In addition, observed case analyses of these assessments at Week 4 and Week 10 were planned.
Time Frame: Visit 1 (Baseline) to Visit 3 (Week 10 or early termination).
Population: This study was terminated early. Secondary efficacy data were not analyzed since only 9 of the 140 planned subjects had been enrolled.
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Donepezil | Placebo
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 1/4 | 3/5
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Donepezil (N=4) | Placebo (N=5)
Bruxism (Gastrointestinal disorders) | 0 | 1
Tongue disorder (Gastrointestinal disorders) | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Abnormal behavior (Psychiatric disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Due to the study terminating early,only 9 subjects were enrolled and these subjects receive only limited exposure to study medications with no subject reaching his/her maximum targeted dose. Therefore,the planned efficacy criteria were not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No